CLINICAL TRIAL: NCT03336229
Title: The Effect of Home-based Prehabilitation on the Cardiorespiratory Fitness of High-risk Colorectal Cancer Patients Awaiting Surgery
Brief Title: Enhancing Fitness With Preoperative Exercise in Colorectal Cancer Surgery
Acronym: EFEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Southampton (Other); NHS Lanarkshire (Other Government); National Heatlh Service Ayrshire and Arran (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GN16OG765
Record Dates: First submitted 2017-09-21; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Cancer
Keywords: cancer; colorectal; exercise; physical fitness
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Exercise intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Exercise intervention — Graduated walking programme, strengthening exercises and respiratory muscle training.
  Arms: Intervention

SUMMARY:
This study examines whether a home-based telephone-guided preoperative exercise programme is feasible and effective in improving cardiorespiratory fitness in patients with colorectal cancer who are high risk due to their existing co-morbidity.

DETAILED DESCRIPTION:
Preoperative exercise, also know as prehabilitation, has been shown to improve physical fitness and potentially reduce postoperative complications in patients undergoing surgery. Patients are often labelled high risk for surgery due to their existing ill-health e.g. heart and lung disease. High risk patients comprise approximately 12% of all elective cancer cases, but account for 80% of all post-operative mortality. Complications significantly affect the quality of life of each CRC patient, both in the short and long-term, and can also impact on survival. It is critical that patients who are deemed at high risk of complications are optimised in the preoperative period. Exercise in the period before surgery is therefore one potential method of improving high risk patients' physical fitness levels while potentially reducing their risk of postoperative complications and subsequent mortality.

ELIGIBILITY:
Inclusion Criteria:

* Primary operable colorectal cancer;
* Awaiting surgery with curative intent;
* Deemed high risk by the responsible clinical team;
* Ability to mobilise independently

Exclusion Criteria:

* Patients with primary or recurrent inoperable colorectal cancer.
* Patients undergoing preoperative chemo- and/or radiotherapy.
* Patients who decline or are deemed unfit for operative management.
* Patients who lack capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Preoperative period: 4 weeks
  Anaerobic threshold as measured by CPET

SECONDARY OUTCOMES:
Length of stay in high dependency and intensive care | Postoperative period: up to 8 weeks
  Critical Care bed days
Readmission to critical care | Postoperative period: up to 8 weeks (within index admission)
  Critical Care bed days
Time to medical discharge | Postoperative period: up to 8 weeks.
  Medically fit for discharge
Hospital length of stay | Postoperative period: within 30 days.
  Days
Readmission rate | Within 30 days of discharge.
Post-operative morbidity | Post-operative period: at 30 days post-surgery (week 8).
  Clavien-Dindo Scale
Health-related quality of life | Baseline (week 0), post-intervention (week 4), at 30 days postoperatively (week 8).
  SF-36
Health-related quality of life | Baseline (week 0), post-intervention (week 4), at 30 days postoperatively (week 8).
  EORTC QLQ-C30
Psychological health | Baseline (week 0), post-intervention (week 4), at 30 days postoperatively (week 8).
  Hospital Anxiety and Depression Score (HADS)
Frailty | Baseline (week 0) and repeat testing (week 4).
  Clinical Frailty Score (CSHA)
Redox blood samples | Baseline (week 0) and repeat CPET (week 4).
  Redox status in pre- and post-exercise blood samples
Survival | 3 years post-operatively.
  Overall and cancer-specific

OTHER OUTCOMES:
Feasibility of home-based exercise | Preoperative period: 4 weeks.
  Recruitment, retention, adherence rates

CONTACTS AND LOCATIONS:
Overall Officials: Katrina A Knight, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (4):
- United Kingdom (4):
  - Hairmyres Hospital, East Kilbride
  - Queen Elizabeth University Hospital, Glasgow
  - University Hospital Crosshouse, Kilmarnock
  - Royal Alexandra Hospital, Paisley

IPD SHARING:
Plan to Share IPD: No